CLINICAL TRIAL: NCT01039077
Title: Single Incision Laparoscopic Gastric Banding Versus Conventional Five Port Laparoscopic Gastric Banding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SLR IRB#08-148
Record Dates: First submitted 2009-12-22; First posted 2009-12-24 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-08

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Single incision laparoscopic gastric banding (Active Comparator): Patients in this group will undergo laparoscopic gastric banding through a single periumbilical incision.
  Interventions: Procedure: Laparoscopic gastric banding
- Five port laparoscopic gastric banding (Active Comparator): Patients in this group will undergo conventional laparoscopic gastric banding using 5 small incisions.
  Interventions: Procedure: Laparoscopic gastric banding

INTERVENTIONS:
Procedure: Laparoscopic gastric banding — Laparoscopic gastric banding for the treatment of morbid obesity.

SUMMARY:
Gastric banding has been shown to significantly reduce weight and has been approved as a treatment of morbid obesity. The standard laparoscopic operation requires five small incisions for the introduction of instruments and the band into the patient's abdomen. We have developed a technique for performing this operation through a single incision at the belly button. This study compares this method to the conventional 5-incision approach.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 40
* ASA Class I or II

Exclusion Criteria:

* Comorbid cardiac, pulmonary, renal, hepatic disease
* Bleeding disorder
* Previous gastric/esophageal surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2009-12; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
weight loss | 1 month and 1 year post-operative

SECONDARY OUTCOMES:
quality of life | 1 week and 3 months post-operative
perioperative complication rate | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Julio Teixeira, MD, Principal Investigator — St. Luke's-Roosevelt Hospital Center
Locations (1):
- St. Luke's-Roosevelt Hospital Center, New York, New York, United States